CLINICAL TRIAL: NCT05035446
Title: A Prospective Randomized Controlled Study of the Short-term Efficacy of Single-hole Plus One-hole Total Laparoscopic Surgery Versus Five-hole Total Laparoscopic Surgery for Distal Gastric Cancer
Brief Title: Short-term Outcomes of SILS+1 Versus CLS for Distal Gastric Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SILS+1-GC-001
Record Dates: First submitted 2021-08-26; First posted 2021-09-05 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-09

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- single-incision plus one-port laparoscopic surgery(SILS + 1) (Experimental): It requires an auxiliary small incision and one more port to perform laparoscopic gastrectomy
  Interventions: Procedure: single-incision plus one-port laparoscopic surgery
- conventional laparoscopic surgery(CLS) (Other): It requires 5 perforations ports and an auxiliary small incision to perform laparoscopic gastrectomy
  Interventions: Procedure: conventional laparoscopic surgery

INTERVENTIONS:
Procedure: single-incision plus one-port laparoscopic surgery — The investigators use the technique of adding one operation hole on the basis of single-port laparoscopy in some patients.
  Arms: single-incision plus one-port laparoscopic surgery(SILS + 1)
Procedure: conventional laparoscopic surgery — It usually requires 5 perforations ports and an auxiliary small incision to perform laparoscopic gastrectomy.
  Arms: conventional laparoscopic surgery(CLS)

SUMMARY:
To evaluate the short-term outcomes of single-incision plus one-port laparoscopic surgery (SILS + 1) versus conventional laparoscopic surgery(CLS) for distal gastric cancer whose clinical stage was cT1-3N0-2M0

DETAILED DESCRIPTION:
The gastric cancer patients with cT1-3N0-2M0 were randomized at a 1:1 ratio to the CLS group or the SILS+1group, then it will evaluate the short-term outcomes between two groups.

ELIGIBILITY:
Inclusion Criteria:

* pathological diagnosis of gastric cancer
* clinically diagnosed cT1b-3N0-2M0 lesions according to the 8th Edition of the American Joint Committee on Cancer(AJCC) Cancer Staging Manual(measured using abdominal CT)
* tumor size ≤ 5cm
* planned to conduct subtotal gastrectomy

Exclusion Criteria:

* preoperative radiotherapy and chemotherapy
* tumor perforation
* severe mental disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Rate of complications | It is within 30 days after surgery
  It means the rate of intraoperative and postoperative complications

SECONDARY OUTCOMES:
Rate of death | It is within 30 days after surgery
  It means the rate of death after operation
pain intensity | 1-3 days after operation
  The investigators use Visual analogue scale(VAS) to evaluate the intensity of pain

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Cancer Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kunisaki C, Miyamoto H, Sato S, Tanaka Y, Sato K, Izumisawa Y, Yukawa N, Kosaka T, Akiyama H, Saigusa Y, Sakamaki K, Yamanaka T, Endo I. Surgical Outcomes of Reduced-Port Laparoscopic Gastrectomy Versus Conventional Laparoscopic Gastrectomy for Gastric Cancer: A Propensity-Matched Retrospective Cohort Study. Ann Surg Oncol. 2018 Nov;25(12):3604-3612. doi: 10.1245/s10434-018-6733-x. Epub 2018 Sep 3. PMID 30178393
- [Background] Kashiwagi H, Kumagai K, Monma E, Nozue M. Dual-port distal gastrectomy for the early gastric cancer. Surg Endosc. 2015 Jun;29(6):1321-6. doi: 10.1007/s00464-014-3827-9. Epub 2014 Aug 27. PMID 25159658
- [Background] Zhou W, Dong CZ, Zang YF, Xue Y, Zhou XG, Wang Y, Ding YL. Initial experience of single-incision plus one port left-side approach totally laparoscopic distal gastrectomy with uncut Roux-en-Y reconstruction. World J Gastroenterol. 2020 Aug 21;26(31):4669-4679. doi: 10.3748/wjg.v26.i31.4669. PMID 32884224
- [Background] Kunisaki C, Makino H, Kimura J, Takagawa R, Ota M, Kosaka T, Akiyama H, Endo I. Application of reduced-port laparoscopic total gastrectomy in gastric cancer preserving the pancreas and spleen. Gastric Cancer. 2015 Oct;18(4):868-75. doi: 10.1007/s10120-014-0441-4. Epub 2014 Nov 15. PMID 25398519
- [Background] Kim SM, Ha MH, Seo JE, Kim JE, Choi MG, Sohn TS, Bae JM, Kim S, Lee JH. Comparison of Reduced Port Totally Laparoscopic Distal Gastrectomy (Duet TLDG) and Conventional Laparoscopic-Assisted Distal Gastrectomy. Ann Surg Oncol. 2015 Aug;22(8):2567-72. doi: 10.1245/s10434-014-4333-y. Epub 2015 Jan 7. PMID 25564174
- [Background] Yang X, Bu Z, He M, Lin Y, Jiang Y, Chen D, Liu K, Zhou J. Effectiveness and safety of reduced-port laparoscopic surgery vs conventional multi-port laparoscopic surgery in the treatment of gastric diseases: A meta-analysis. Medicine (Baltimore). 2021 Jan 22;100(3):e23941. doi: 10.1097/MD.0000000000023941. PMID 33545969
- [Background] Kim SM, Ha MH, Seo JE, Kim JE, Choi MG, Sohn TS, Bae JM, Kim S, Lee JH. Comparison of single-port and reduced-port totally laparoscopic distal gastrectomy for patients with early gastric cancer. Surg Endosc. 2016 Sep;30(9):3950-7. doi: 10.1007/s00464-015-4706-8. Epub 2015 Dec 22. PMID 26694180
- [Background] Kim HG, Kim DY, Jeong O. Transition from Conventional to Reduced-Port Laparoscopic Gastrectomy to Treat Gastric Carcinoma: a Single Surgeon's Experience from a Small-Volume Center. J Gastric Cancer. 2018 Jun;18(2):172-181. doi: 10.5230/jgc.2018.18.e18. Epub 2018 Jun 27. PMID 29984067
- [Background] Lu YM, Lin T, Hu YF, Liu H, Mou TY, Zhu Y, Yu J, Li GX. Initial Experience of Dual-Port Laparoscopic Distal Gastrectomy for Gastric Cancer: A Single-Arm Study. Adv Ther. 2019 Sep;36(9):2342-2350. doi: 10.1007/s12325-019-01029-x. Epub 2019 Jul 23. PMID 31338689